CLINICAL TRIAL: NCT01182688
Title: Prospective Review of Procalcitonin After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Tampa Bay Heart Foundation (Other)
Responsible Party: Devednra Amin, MD, Bay Area Chest Physicians, PA
Other Study IDs: 2008.023; 2008.023 (Other Grant/Funding Number: TampaBay Heart Foundation)
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2009-10

CONDITIONS: Procalcitonin; Coronary Artery Bypass Grafting
Keywords: utilization of Procalcitonin in the cardiac setting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to demonstrate the value of Procalcitonin (PCT) in assisting the rapid diagnosis of post- operative infection that includes elevation of Procalcitonin above and beyond the changes seen with the acute and inflammatory response induced by cardio-pulmonary bypass.

Procalcitonin is an innovative and highly specific biomarker for clinically relevant severe bacterial infections and sepsis. PCT supports early diagnosis and clinical decision making.This is a prospective single center study designed to assess the normal change in PCT levels following major surgery and the utilization of PCT regarding the diagnosis of infection and the response to treatment, following major cardiac surgery

DETAILED DESCRIPTION:
Inclusion Criteria:

Elective CABG + / - Aortic / Mitral valve patients Off pump and on pump cases

Exclusion Criteria:

Patients with recent infection in last week and / or Antibiotics in last 1 week or pre op fever > 99.5f / 38C in 24hrs prior to surgery Patients on oral or IV corticosteroids within 1 week of being on them. Known immune dysfunction Active congestive heart failure / Recovering from cardiogenic shock\ Intra aortic balloon pump pre - op No CABG patients with CRYO MAZE, or Ablation

ELIGIBILITY:
Inclusion Criteria:

Elective CABG + / - Aortic / Mitral valve patients Off pump and on pump cases

Exclusion Criteria:

Exclusion Criteria:

Check any box that applies:

Patients with recent infection in last week and / or Antibiotics in last 1 week or pre op fever > 99.5f / 38C in 24hrs prior to surgery Patients on oral or IV corticosteroids within 1 week of being on them. Known immune dysfunction Active congestive heart failure / Recovering from cardiogenic shock\ Intra aortic balloon pump pre - op No CABG patients with CRYO MAZE, or Ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having Elective CABG + / - Aortic / Mitral valve patients Off pump and on pump cases
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Morton Plant Hospital, Clearwater, Florida, United States